CLINICAL TRIAL: NCT06379919
Title: Cutibacterium Acnes Removal by Wound Irrigation With Normal Saline Versus Irrisept During Total Shoulder Arthroplasty
Brief Title: Wound Irrigation Comparative Effectiveness Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopaedic Education and Research Institute (dba Hoag Orthopedics) (Other)
Collaborators: Irrimax Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C Acnes in TSA
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Cutibacterium Acnes Contamination

STUDY DESIGN:
Intervention Model Description: Participants are assigned at the beginning of the study to treatment arm involving 1 of 2 types of irrigation treatment for their surgery. They continue in that arm through the length of the study and complete the same study procedures, as well as same standard of care.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and Microbiology lab assessing cultures are blinded to the assigned irrigation treatment arm throughout the length of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline Irrigation Arm (Group 1) (Active Comparator): After deep dissection, and prior to implantation of components, 100 cc of normal saline will be irrigated into the deep wound and progress outward through more superficial planes to the skin. Cultures will then be taken at multiple wound depths and time points.
  Interventions: Procedure: Saline Irrigation Solution Delivery
- Irrisept irrigation Arm (Group 2) (Active Comparator): After deep dissection, and prior to implantation of components, 100 cc of Irrisept solution will be irrigated into the deep wound and progress outward through more superficial planes to the skin. Cultures will then be taken at multiple wound depths and time points.
  Interventions: Procedure: Irrisept Irrigation

INTERVENTIONS:
Procedure: Irrisept Irrigation — Irrisept Antimicrobial Wound Lavage is a single-use, manual, self-contained irrigation device. Irrisept contains 0.05% Chlorhexidine Gluconate (CHG) in 99.95% Sterile Water for Irrigation, United Staes Pharmacopeia (USP). The solution is aseptically filled in a Blow-Fill-Seal (BFS) bottle.
  Other Names: Chlorohexidine Gluconate Solution Delivery
  Arms: Irrisept irrigation Arm (Group 2)
Procedure: Saline Irrigation Solution Delivery — Normal saline is isotonic and the most commonly used wound irrigation solution due to safety (lowest toxicity) and physiologic factors.
  Arms: Normal Saline Irrigation Arm (Group 1)

SUMMARY:
The primary objective of this study is to compare the presence of C acnes in bacteriologic cultures taken from participant samples of subcutaneous and deep tissue prior to deep surgical irrigation using either Normal Saline Irrigation (Group 1) or Irrisept Irrigation (Group 2). Secondary objectives are evaluation of patient reported outcome measures and range of motion in relation to C acnes presence among subjects in the two groups.

ELIGIBILITY:
Inclusion Criteria:

• Ault patients requiring Total Shoulder Arthroplasty

Exclusion Criteria:

* Age younger than 18 years
* History of shoulder infection
* Antibiotic therapy within 2 weeks of surgery
* Cortisone infiltration within 3 months prior to surgery
* Allergy to CHG
* Diagnosis of rheumatoid arthritis
* Immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
C Acnes Presence | Cultures take during surgery and analyzed over 21 days post surgery
  The primary outcome of this study is to compare the presence of C acnes in bacteriologic cultures taken from participant samples of subcutaneous and deep tissue prior to deep surgical irrigation using either Normal Saline Irrigation (Group 1) or Irrisept Irrigation (Group 2)rimary objecti

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Patient Reported Outcome Measure | Pre-operation, 3, 6, 12, & 24 Months post-operation,
  This assessment consists of 17, multiple choice questions that pertain to pain and function of the operated shoulder.
Shoulder Range of Motion (ROM) | Pre-operation, 3, 6, 12, & 24 Months post-operation,
  Shoulder Range of Motion will require the Investigator or Designee to evaluate the following degrees of freedom:
  Forward flexion
  External Rotation with elbow at side
  External Rotation with elbow at 900
  Internal Rotation as measured by spinal segment reached.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiz F Kassam, MD, Principal Investigator — Hoag Orthopedics Education and Research
Locations (1):
- Hoag Orthopedics, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Athwal GS, Sperling JW, Rispoli DM, Cofield RH. Deep infection after rotator cuff repair. J Shoulder Elbow Surg. 2007 May-Jun;16(3):306-11. doi: 10.1016/j.jse.2006.05.013. Epub 2007 Feb 22. PMID 17321157
- [Background] Horneff JG 3rd, Hsu JE, Voleti PB, O'Donnell J, Huffman GR. Propionibacterium acnes infection in shoulder arthroscopy patients with postoperative pain. J Shoulder Elbow Surg. 2015 Jun;24(6):838-43. doi: 10.1016/j.jse.2015.03.008. PMID 25979553
- [Background] Foster AL, Cutbush K, Ezure Y, Schuetz MA, Crawford R, Paterson DL. Cutibacterium acnes in shoulder surgery: a scoping review of strategies for prevention, diagnosis, and treatment. J Shoulder Elbow Surg. 2021 Jun;30(6):1410-1422. doi: 10.1016/j.jse.2020.11.011. Epub 2020 Dec 26. PMID 33373684
- [Background] Chuang MJ, Jancosko JJ, Mendoza V, Nottage WM. The Incidence of Propionibacterium acnes in Shoulder Arthroscopy. Arthroscopy. 2015 Sep;31(9):1702-7. doi: 10.1016/j.arthro.2015.01.029. Epub 2015 Mar 29. PMID 25823673
- [Background] Dizay HH, Lau DG, Nottage WM. Benzoyl peroxide and clindamycin topical skin preparation decreases Propionibacterium acnes colonization in shoulder arthroscopy. J Shoulder Elbow Surg. 2017 Jul;26(7):1190-1195. doi: 10.1016/j.jse.2017.03.003. Epub 2017 May 4. PMID 28479255
- [Background] Millett PJ, Yen YM, Price CS, Horan MP, van der Meijden OA, Elser F. Propionibacterium acnes infection as an occult cause of postoperative shoulder pain: a case series. Clin Orthop Relat Res. 2011 Oct;469(10):2824-30. doi: 10.1007/s11999-011-1767-4. Epub 2011 Jan 15. PMID 21240577
- [Background] Contreras ES, Frantz TL, Bishop JY, Cvetanovich GL. Periprosthetic Infection After Reverse Shoulder Arthroplasty: a Review. Curr Rev Musculoskelet Med. 2020 Dec;13(6):757-768. doi: 10.1007/s12178-020-09670-8. PMID 32827305
- [Background] Cooper ME, Trivedi NN, Sivasundaram L, Karns MR, Voos JE, Gillespie RJ. Diagnosis and Management of Periprosthetic Joint Infection After Shoulder Arthroplasty. JBJS Rev. 2019 Jul;7(7):e3. doi: 10.2106/JBJS.RVW.18.00152. No abstract available. PMID 31291202
- [Background] Lemmens L, Geelen H, Depypere M, De Munter P, Verhaegen F, Zimmerli W, Nijs S, Debeer P, Metsemakers WJ. Management of periprosthetic infection after reverse shoulder arthroplasty. J Shoulder Elbow Surg. 2021 Nov;30(11):2514-2522. doi: 10.1016/j.jse.2021.04.014. Epub 2021 Apr 22. PMID 33895302
- [Background] Horneff JG, Hsu JE, Huffman GR. Propionibacterium acnes infections in shoulder surgery. Orthop Clin North Am. 2014 Oct;45(4):515-21. doi: 10.1016/j.ocl.2014.06.004. Epub 2014 Jul 11. PMID 25199422
- [Background] Heckmann N, Heidari KS, Jalali O, Weber AE, She R, Omid R, Vangsness CT, Rick Hatch GF 3rd. Cutibacterium acnes persists despite topical clindamycin and benzoyl peroxide. J Shoulder Elbow Surg. 2019 Dec;28(12):2279-2283. doi: 10.1016/j.jse.2019.06.016. Epub 2019 Aug 27. PMID 31471244
- [Background] Phadnis J, Gordon D, Krishnan J, Bain GI. Frequent isolation of Propionibacterium acnes from the shoulder dermis despite skin preparation and prophylactic antibiotics. J Shoulder Elbow Surg. 2016 Feb;25(2):304-10. doi: 10.1016/j.jse.2015.08.002. Epub 2015 Oct 9. PMID 26456428
- [Background] McDonnell G, Russell AD. Antiseptics and disinfectants: activity, action, and resistance. Clin Microbiol Rev. 1999 Jan;12(1):147-79. doi: 10.1128/CMR.12.1.147. PMID 9880479
- [Background] Edmiston CE Jr, Bruden B, Rucinski MC, Henen C, Graham MB, Lewis BL. Reducing the risk of surgical site infections: does chlorhexidine gluconate provide a risk reduction benefit? Am J Infect Control. 2013 May;41(5 Suppl):S49-55. doi: 10.1016/j.ajic.2012.10.030. PMID 23622749
- [Background] Falconer TM, Baba M, Kruse LM, Dorrestijn O, Donaldson MJ, Smith MM, Figtree MC, Hudson BJ, Cass B, Young AA. Contamination of the Surgical Field with Propionibacterium acnes in Primary Shoulder Arthroplasty. J Bone Joint Surg Am. 2016 Oct 19;98(20):1722-1728. doi: 10.2106/JBJS.15.01133. PMID 27869623
- [Background] Moor BK, Leger B, Steffen V, Troillet N, Emonet S, Gallusser N. Subcutaneous tissue disinfection significantly reduces Cutibacterium acnes burden in primary open shoulder surgery. J Shoulder Elbow Surg. 2021 Jul;30(7):1537-1543. doi: 10.1016/j.jse.2020.11.018. Epub 2021 Jan 6. PMID 33421560
- [Background] Hudek R, Brobeil A, Bruggemann H, Sommer F, Gattenlohner S, Gohlke F. Cutibacterium acnes is an intracellular and intra-articular commensal of the human shoulder joint. J Shoulder Elbow Surg. 2021 Jan;30(1):16-26. doi: 10.1016/j.jse.2020.04.020. Epub 2020 Jun 9. PMID 32741563